CLINICAL TRIAL: NCT06602895
Title: Shaping Champions: a Cutting-Edge Analysis of Physical Performance in Male and Female National Kho-Kho Players Following Intensive Functional Training
Brief Title: Assessing Physical Performance in Male and Female National Kho-Kho Players Following Intensive Functional Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRIIRS/FAHS/DEC/2021-S006
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Physical Performance
Keywords: Agility; Functional performance; Kho-Kho; Static Balance; Dynamic balance

STUDY DESIGN:
Intervention Model Description: pretest-posttest gender-based parallel group comparative design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Male group (Active Comparator): The male group received intensive short-term functional strength training and balance training consecutively for one hour each, six days a week for two weeks.
  Interventions: Other: Intensive short-term functional strength training; Other: Balance Training
- Female group (Active Comparator): The female group received balance training and intensive short-term functional strength training consecutively for one hour each, six days a week for two weeks.
  Interventions: Other: Intensive short-term functional strength training; Other: Balance Training

INTERVENTIONS:
Other: Intensive short-term functional strength training — All players underwent a rigorous 2-week intensive short-term functional strength training program, with training sessions held for 5 days a week. One group engaged in intensive short-term functional strength training exercises, while the other group focused on balance training. The training regimen was then reversed for the two groups. Each daily training session lasted approximately 2 hours, with 1 hour of either intensive short-term functional strength training or balance training. Every intensive short-term functional strength training session spanned roughly 60 minutes, starting with a 10-minute warm-up followed by dynamic mobility exercises targeting key joints. During the 40-minute core segment of our intensive short-term functional strength training sessions, participants first engaged in stability exercises for 10 minutes, focusing on core stability and balance through plank variations and stability.
Other: Balance Training — Participants first engaged in stability exercises for 10 minutes, focusing on core stability and balance through plank variations and stability ball exercises. This was followed by 15 minutes of multi-joint strength exercises, where athletes performed compound movements like squats, deadlifts, push-ups or bench presses, and pull-ups or lat pull-downs, each for t sets of 8-10 repetitions. The session concluded with 15 minutes of agility and coordination drills, incorporating high-intensity activities such as lateral sprints and rope pulling, specifically designed to improve quickness and neuromuscular coordination, thereby enhancing overall athletic performance. The session concluded with a 10-minute cooldown involving flexibility exercises for the limbs and trunk. Exercise intensity was regulated to correspond with a 6-7 on the repetitions in the reserve-based Rating of Perceived Exertion (RPE) scale, where a s indicates that the exerciser feels they could perform approximately.

SUMMARY:
This clinical trial aims to learn if intensive short-term functional strength training works to improve agility, functional movement, and balance among male and female national Kho-Kho players. It will also teach about the effect of gender on physical performance. The main questions it aims to answer are:

* Does the intensive short-term functional strength training work to improve agility, functional movement, and balance among male and female national Kho-Kho players?
* Which gender brings the greater impact on the physical performance of national Kho-Kho players? Researchers will investigate the impact of intensive short-term functional strength training on agility, functional movement, and balance among male and female national Kho-Kho players and compare the impact of male and female differences on physical performance.

Participants will:

• Both male and female groups of participants received an application of intensive short-term functional strength training and balance training or balance training and intensive short-term functional strength training consecutively for one hour each, six days a week for two weeks.

DETAILED DESCRIPTION:
Kho-Kho and kabaddi are two of the most beloved team sports in rural India, and they are celebrated for their historical roots. As Indigenous games of India, they stand out for requiring players to evade contact with opponents. These games are highly competitive, starting from the elementary level and continuing to the national stage, driving both enthusiasm and rivalry. Playing Kho-Kho not only improves physical fitness but also positively impacts mental health, stress management, and overall well-being, contributing to high performance in sports. Notably, adolescent girls face distinct biomechanical and anatomical challenges in Kho-Kho. Functional Strength Training (FST), a comprehensive method, improves athletes' movement efficiency by engaging multiple muscle groups across different planes, making it ideal for improving athletic performance. Intensive FST is essential for optimizing athlete readiness, offering valuable insights to both scientists and coaches on the effectiveness of training programs.

ELIGIBILITY:
Inclusion Criteria:

* Kho-Kho players aged between 18 and 25 years, all at the national level.
* Both male and female participants.
* Expressed eagerness to participate in the camp and training.
* Participants needed foundational experience with functional training relevant to Kho-Kho to ensure they could safely engage in and benefit from the specific training protocols designed for this study.

Exclusion Criteria:

* The participants were unable to perform the required tests and training sessions at the outset.
* Participants with a history of serious injuries related to strength and balance training were also excluded to minimize the risk of re-injury.
* Participants who experienced issues such as low back pain, vestibular problems, or lower extremity injuries during the camp training were removed from the final analysis to ensure the accuracy and integrity of the study's results

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male and Female
Enrollment: 60 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen (FMS) | 2weeks
  The Functional Movement Screen (FMS) is a screening tool that consists of seven motor tasks, encompassing overhead squats, inline lunges, step downs, shoulder flexibility, straight leg lifts, trunk stability pushups, and pushups. Each task is assessed using a conventional 0-3 ordinal system.
  A score of 3 indicates correct execution without pain or compensatory movements, a score of 2 indicates compensatory movements were observed, a score of 1 signifies an inability to complete the movement, and a score of 0 implies no pain during the movement.
  Each exercise is repeated three times, and the best performance is recorded.
  The FMS yields a maximum score of 21, with a total score of 14 or below indicating a higher risk of sports injury development.

SECONDARY OUTCOMES:
Balance | 2weeks
  For the balance study, a biomechanical examination of stability was conducted. Tecnobody, Italy, Prokin 252 N system, was employed to assess both static and dynamic stability components.
  To evaluate static stability, stabilometric tests were performed with both open and closed eyes. To determine dynamic stability balance, the Stability Index was assessed while participants stood on one foot (in the Romberg position) and both feet (in the sharpened Romberg posture).
  Postural sway in degrees was measured for both static and dynamic balance.

OTHER OUTCOMES:
Agility | 2weeks
  The players performed three types of agility tests: the SEMO test, the 40-meter run test, and the Illinois agility test.
  The SEMO Agility Test was conducted following the procedures outlined in a previous study. It measures running agility, incorporating movements such as running backwards and sideways.
  In the 40-meter run test for agility, the players ran as fast as possible between two parallel lines spanning 40 meters.
  Last, the Illinois agility test required athletes to exhibit acceleration, deceleration, and quick changes in direction around numerous cones, completing 90-180-degree revolutions over a 60-meter distance.

CONTACTS AND LOCATIONS:
Overall Officials: Moattar R. Rizvi, PhD, Principal Investigator — Department of Physiotherapy, Manav Rachna International Institute and Studies, Faridabad, India
Locations (1):
- Manav Rachna Sports Science Center, Faridabad, Haryana, India